CLINICAL TRIAL: NCT02920775
Title: Monitoring Patterns of Prescribing to Identify Changes in Access to ER/LA Opioid Analgesics
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ER/LA Opioid REMS Program Companies (RPC) (Industry)
Responsible Party: Sponsor
Other Study IDs: Assessment 8
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Opioid Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (15):
- Pain
  Interventions: Other: Non-interventional study - retrospective database review
- PCP
  Interventions: Other: Non-interventional study - retrospective database review
- Dentist
  Interventions: Other: Non-interventional study - retrospective database review
- Surgery
  Interventions: Other: Non-interventional study - retrospective database review
- Emergency Medicine
  Interventions: Other: Non-interventional study - retrospective database review
- Oncology
  Interventions: Other: Non-interventional study - retrospective database review
- Hospice and Palliative Medicine
  Interventions: Other: Non-interventional study - retrospective database review
- Anesthesiology
  Interventions: Other: Non-interventional study - retrospective database review
- Neurology
  Interventions: Other: Non-interventional study - retrospective database review
- Nurse Practitioners
  Interventions: Other: Non-interventional study - retrospective database review
- Pediatrics
  Interventions: Other: Non-interventional study - retrospective database review
- Physical Medicine & Rehabilitation
  Interventions: Other: Non-interventional study - retrospective database review
- Physician Assistant
  Interventions: Other: Non-interventional study - retrospective database review
- Rheumatology
  Interventions: Other: Non-interventional study - retrospective database review
- All Other Specialties
  Interventions: Other: Non-interventional study - retrospective database review

INTERVENTIONS:
Other: Non-interventional study - retrospective database review

SUMMARY:
Changes in prescribing will be compared in prescribers from specialties whose prescribing is hypothesized to be relatively unaffected by the REMS (such as oncologists and hospice providers) versus those for whom the REMS could have greater impact on prescribing (e.g., dentists). Trends and changes in monthly prescription volume and average monthly prescription volume will be evaluated by prescriber specialty.

ELIGIBILITY:
Inclusion Criteria:

* Changes in number of prescriptions for prescriber types with less or more compelling reasons to prescriber ER/LA opioid analgesics

Exclusion Criteria:

* None

Max Age: 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects filling a prescription for a product of interest as gathered from the IMS National prescription Audit™ and IMS Health, LifeLink™
Sampling Method: Non-Probability Sample
Enrollment: 360000 (Estimated)
Dates: Primary Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Monthly volume of prescriptions by specialty | July 2010-December 2014